CLINICAL TRIAL: NCT06359925
Title: Comparative Study Between Dexmedetomidine Plus Bupivacaine Versus Bupivacaine in Suprazygomatic Maxillary Nerve Block for Management of Postoperative Pain in Tonsillectomy Patients.
Brief Title: Suprazygomatic Nerve Block in Tonsillectomy Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Asaad Hasan Rizk, Assistant Lecturer, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Suprazygomatic nerve block
Record Dates: First submitted 2024-03-22; First posted 2024-04-11 (Actual); Last update posted 2024-04-11 (Actual); Status verified 2024-04

CONDITIONS: Tonsillectomy
MeSH Terms: interventions — Bupivacaine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group S (Active Comparator): Suprazygomatic maxillary nerve block using Dexmedetomidine Plus Bupivacaine
  Interventions: Procedure: Suprazygomatic maxillary nerve block using dexmedetomidne and Bupivacaine
- Group c( control) (Placebo Comparator): Suprazygomatic maxillary nerve block using Bupivacaine only
  Interventions: Procedure: Suprazygomatic maxillary nerve block using Bupivacaine

INTERVENTIONS:
Procedure: Suprazygomatic maxillary nerve block using dexmedetomidne and Bupivacaine — After induction of general anaesthesia blockade of the contents of the pterygopalatine fossa is performed bilaterally before starting surgery as follows: After complete aseptic skin preparation and under ultrasound guidance images are obtained with a high-frequency linear array probe. The ultrasound transducer is placed in the infrazygomatic area, over the maxilla, angled [45 ]degree cephalad. This probe position allows visualization of the pterygopalatine fossa,The needle is advanced using an out-of-plane approach, and the needle tip can usually be identified during movements. the injectate consisted of [4]mL of [0.5% ]Bupivacaine combined with [1]mL of[ 5]µg dexmedetomidine. The injectate is delivered over [15-20 ] seconds, while observing the spread of the local anesthetic under ultrasoundThe same procedure is then repeated on the contralateral side.
  Arms: Group S
Procedure: Suprazygomatic maxillary nerve block using Bupivacaine — After induction of general anaesthesia blockade of the contents of the pterygopalatine fossa is performed bilaterally before starting surgery as follows: After complete aseptic skin preparation and under ultrasound guidance images are obtained with a high-frequency linear array probe. The ultrasound transducer is placed in the infrazygomatic area, over the maxilla, angled [45 ]degree cephalad. This probe position allows visualization of the pterygopalatine fossa,The needle is advanced using an out-of-plane approach, and the needle tip can usually be identified during movements. the injectate consisted of [4]mL of [0.5% ]Bupivacaine combined with [1]mL normal saline . The injectate is delivered over [15-20 ] seconds, while observing the spread of the local anesthetic under ultrasoundThe same procedure is then repeated on the contralateral side.
  Arms: Group c( control)

SUMMARY:
The use of suprazygomatic maxillary nerve block to reduce postoperative pain and hospital stay is greater than the use of NSAID and opioids.

DETAILED DESCRIPTION:
Tonsillectomy is one of the most commonly performed operations worldwide, with postoperative pain being the main cause of morbidity . Unlike most other surgeries, tonsillectomies leave an open wound that heals by secondary intention. Thermal and mechanical injuries lead to inflammation, nerve irritation, and spasms of the pharyngeal muscles that can result in severe pain Because, this procedure is performed primarily on an outpatient basis, postoperative complications, including pain, vomiting, fever, and hemorrhage, can significantly lengthen recovery room stays and lead to emergency department visits and unanticipated hospital admission.

Poorly controlled posttonsillectomy pain can result in decreased oral intake, dysphagia, dehydration, and weight loss. Standard management of postoperative pain following tonsillectomy includes acetaminophen, hydrocodone or oxycodone, and nonsteroidal anti-inflammatory drugs .

Despite scheduled administration of analgesics, postoperative pain is often poorly controlled .

Opioid use and preoperative pain at or remote from the surgical site have been demonstrated to be associated with a higher risk of persistent postoperative pain ,and large cohort studies have reported concerning rates of long-term postoperative opioid use after minor surgery in previously opioid-naı¨ve patients .

Efforts to reduce opioid use, particularly after hospital discharge, require further attention; thus opioid consumption beyond the early postoperative period is an increasingly important outcome measure .

As systemic analgesics have proven inefficacious and insufficient to reliably control post-tonsillectomy pain, regional anesthetic techniques are an option, and although they are in their infancy in terms of development and rarely utilized, they may offer advantages over standard approaches. The tonsils are innervated both by branches of the maxillary division of the trigeminal nerve via the lesser (and perhaps greater) palatine nerves and the tonsillar branches of the glossopharyngeal nerve, whereas the adenoids are innervated exclusively by branches of the lesser palatine nerve. Although some studies have indicated significant reduction of postoperative pain with both pre-incisional ropivacaine injected into the tonsillar fossa and postincisional topical ropivacaine in the tonsillar fossa, a Cochrane review of local anesthetics to reduce post-tonsillectomy pain found no evidence of efficacy .

Given the insufficient evidence and risk of inadvertent injection into the carotid artery, the use of local anesthetics at the surgical site is not currently recommended .

Local anesthetic injected into the pterygopalatine fossa has been described for pediatric cleft palate repair with excellent control of postoperative pain compared with systemic analgesics .

The need for postoperative morphine was completely eradicated in one study. The effects of local anesthetic have been noted to have effects on pain for an inexplicably long period (up to 10 days after injection), long after the local anesthetic wears off The tonsillar bed is innervated by the lesser (and perhaps greater) palatine nerve and the glossopharyngeal nerve . Given that both the greater and lesser palatine nerves originate in the pterygopalatine fossa, this space is a logical anatomic target for regional anesthesia to cover the tonsillar fossa .Targeting of the glossopharyngeal nerve for blockade, while possible, would also ablate the gag reflex, which carries an unacceptably high risk of airway compromise in the aftermath of pharyngeal surgery. The suprazygomatic approach to the pterygopalatine fossa is a technically easy procedure to perform with ultrasound guidance, with an average procedure time of 56 seconds . Suprazygomatic approaches to the pterygopalatine fossa have been associated with fewer complications than infrazygomatic approaches, which include orbital puncture, intracranial injection, maxillary artery puncture, or posterior pharyngeal wall injury .

Using a suprazygomatic approach and ultrasound guidance, Sola et al. experienced zero technical complications after 50 blocks

ELIGIBILITY:
Inclusion Criteria:

* Children aged 3-10 years old
* The American Society of Anesthesiologists (ASA) I and II
* Children scheduled for tonsillectomy with or without adenoidectomy.

Exclusion Criteria:

* Patient's guardian refusal to participate in the study.
* Children with Behavioural changes; physical or developmental delay; neurological disorder or psychological disorder.
* Children on sedative or anticonvulsant medication.
* Bleeding diathesis
* History of sleep apnea
* Significant organ dysfunction.
* cardiac dysrhythmia.
* congenital heart disease .
* Known allergy to the study drugs.
* Skin lesions or wounds at the puncture site of the proposed block

Ages: 3 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2024-10-22 (Estimated); Primary Completion 2025-09-20 (Estimated); Study Completion 2026-02-20 (Estimated)

PRIMARY OUTCOMES:
time and amount of first postoperative rescue analgesia after two different blocks using Children's Hospital of Eastern Ontario Pain Scale (CHEOPS) score | 24 hours
  Postoperative pain will be recorded using Children's Hospital of Eastern Ontario Pain Scale (CHEOPS) scores at admission to the PACU [0] minutes (baseline), [30 ]minutes, [1], [4], [8],[ 12], [18] and [24] hours postoperatively. where the minimum score of zero (no pain) and the maximum score of 12 (the most severe pain). Children with the modified CHEOPS [ ≥ 5 ]will be given supplemental analgesia with IV paracetamol 15 mg/kg , Pain scores will be recorded 15-20 minutes following the administration of this supplemental analgesia to assess pain relief. The number of children that required postoperative rescue analgesics, the first time to rescue analgesia, and the total amount of rescue analgesia consumed within [24] hours postoperatively will be recorded.

SECONDARY OUTCOMES:
time and amount of first postoperative rescue analgesia after two different blocks using Paediatric Anaesthesia Emergence Delirium (PAED) scale | 24 hours
  Emergency agitation (EA) will be evaluated using Paediatric Anaesthesia Emergence Delirium (PAED) scale; upon admission to the PACU (0 min, baseline),( 30), and( 60 ) min until discharge from the PACU.
  The highest EA scores observed during this period will be recorded. PAED score ≥ 10 will be considered to be a diagnostic endpoint for the development of agitation.
  Emergence agitation and postoperative pain (scores of ≥ 10) will be managed by intravenous doses of fentanyl( 0.5) mic/kg, repeated after [10 ] min if the child still agitated or in pain, with a maximum total dose of 2 mic/kg. Patients who showed EA were monitored continuously until the EA subsided spontaneously or with medication.
Parents satisfaction score | 24 hours
  Parental satisfaction will be determined 24 h after the surgery by an anesthetist blinded to the study groups. The child's comfort, activity level and the presence or absence of pain will be used to determine the result as 1 (unsatisfied), 2 (satisfied or good), or 3 (very satisfied or excellent)